CLINICAL TRIAL: NCT01907841
Title: The Effect of Ischemic Pre-Conditioning on the Rate of Recovery Following Exercise-Induced Muscle Damage: a Randomized Control Trial
Brief Title: The Effect of Ischemic Pre-Conditioning on the Rate of Recovery Following Exercise-Induced Muscle Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Mary's University College (Other)
Responsible Party: Principal Investigator, Stephen Patterson, Senior Lecturer Exercise Physiology, St Mary's University College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPCEIMD001
Record Dates: First submitted 2013-07-15; First posted 2013-07-25 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Exercise-induced Muscle Damage
Keywords: Investigate IPC on EIMD
MeSH Terms: interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ischemic Preconditioning (Experimental): IPC (4 x 5 minute cycles @ 220 mmHg) with 5 min reperfusion between trials.
  Interventions: Other: Ischemic Preconditioning
- Ischemic Preconditioning Placebo (Placebo Comparator): Placebo (4 x 5 minute cycles @ 20mmHg) with 5 minutes between each cycle
  Interventions: Other: Ischemic Preconditioning

INTERVENTIONS:
Other: Ischemic Preconditioning

SUMMARY:
Strenuous exercise or exercise involving eccentric muscle contractions can lead to muscle damage and changes in muscle function; this is known as exercise-induced muscle damage (EIMD). It is known that brief, repeated periods of ischemia followed by reperfusion, known as Ischemic Preconditioning (IPC) cause a delay in cell injury in cardiac muscle as well as in various other organs.

Therefore the purpose of this study is to:

1. Quantify the use of IPC in recovery following EIMD.
2. Identify any effect of IPC during recovery on muscle function

ELIGIBILITY:
Inclusion Criteria:

* Physically Active Males

Exclusion Criteria:

* Muscular skeletal disorders

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in maximal voluntary contraction | pre exercise, 24 hours post, 48 hours post and 72 hours post exercise
  Isometric MVC of the participants' dominant knee extensors was assessed using a strain gauge. MVCs were performed for 3 s with a 60 s rest between each repetition.
  The change in MVC will be determined 24, 48 and 72 hours following pre exercise conditions.

SECONDARY OUTCOMES:
Change from baseline in Creatine kinase | pre exercise, 24 hours post, 48 hours post and 72 hours post exercise
  Plasma CK was determined from an earlobe capillary blood sample. The sample (10 microlitres) was analysed immediately using an semi-automated clinical chemistry analyser.
  The change in CK will be determined 24, 48 and 72 hours following pre exercise conditions
Change from baseline in Limb girth | pre exercise, 24 hours post, 48 hours post and 72 hours post exercise
  Mid-thigh and calf circumference was assessed as a measure of limb swelling using an anthropometric tape measure. Both measures were obtained with the participant in a standing position.
  The change in limb girth will be determined 24, 48 and 72 hours following pre exercise conditions
Chnage from baseline in Vertical jump | pre exercise, 24 hours post, 48 hours post and 72 hours post exercise
  Vertical jump (VJ) performance was assessed using an electronic timing mat with hands placed on hips and participants dropping down to a self-selected level before jumping maximally.
  The change in VJ will be determined 24, 48 and 72 hours following pre exercise conditions
Change from baseline in Muscle soreness | pre exercise, 24 hours post, 48 hours post and 72 hours post exercise
  Muscle soreness - Participants were asked to perform and hold a squat (90° knee angle) whilst they rated their perceived muscle soreness on a 200 mm visual analogue scale. The scale consisted of a line from 0 mm (no pain) to 200 mm (unbearably painful).
  The change in muscle soreness will be determined 24, 48 and 72 hours following pre exercise conditions

CONTACTS AND LOCATIONS:
Locations (1):
- St Marys Umiversity College, London, United Kingdom